CLINICAL TRIAL: NCT05448586
Title: Opioid Free Anaesthesia in Oncologic Gynaecological Surgery: Is There Any Benefit? Retrospective Observational Study
Brief Title: Opioid Free Anaesthesia in Oncologic Gynaecological Surgery: Is There Any Benefit?
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: PI-3958
Record Dates: First submitted 2022-01-12; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2021-02

CONDITIONS: Cervix Cancer; Endometrial Cancer; Ovarian Cancer; Breast Cancer
Keywords: Opioid; Opioid Free Anesthesia; SIRS (Systemic Inflammatory Response); Postoperative infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Breast Neoplasms | interventions — Analgesics, Opioid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Balanced anesthesia with opioids: Patients who had Major Surgery for gynecologic cancers (cervix, endometrium, ovarian and breast cancer) under balanced anesthesia including opioids between February 2019 and 2020 in Hospital La Paz.
  Interventions: Drug: Opioid
- Opioid Free Anesthesia (OFA): Patients who had Major Surgery for gynecologic cancers (cervix, endometrium, ovarian and breast cancer) under Opioid Free anesthesia between February 2019 and 2020 in Hospital La Paz.

INTERVENTIONS:
Drug: Opioid — Use of balanced anesthesia including opioids during anesthesia for gynecologic cancer surgery
  Other Names: Opioid Free Anesthesia
  Groups: Balanced anesthesia with opioids

SUMMARY:
Opioid Free Anesthesia (OFA) is a multimodal anesthesia and emerging technique that spares the use of opioids and involve other adjuvant anesthetics, which have demonstrated in vitro influence on immunologic and inflammatory response, as well as in metastatic progression. For these reasons we believe that OFA may positively influence in oncologic patients postoperative recovery and in its disease progression.

DETAILED DESCRIPTION:
After Local Ethics Committee approval, consecutive consenting patients scheduled for major gynecologic oncologic surgery were included between February 2019 and January 2020 in this observational retrospective study. We Compared OFA to standard technique used in our institution and assessed its effect on Postoperative Systemic Inflammatory Response (SIRS), hospital stay, postoperative complications in the following 2 months, cancer progression and mortality 6 months and 12 months after surgery. OFA protocol consisted of a Total IntraVenous Anaesthesia of Propofol, a Dexmedetomidine infusion of 0,8-1,0 mcg/kg/h, together with 0,2-0,3 mg/kg ketamine and lidocaine 1,5 mg/kg in the first hour of surgery. The standard anaesthetic protocol included opioids (Fentanyl 2mcg/kg at induction, and remifentanyl infusion 0,1-0,2 mcg/kg/min) and volatile agents (sevoflurane or desflurane). Patients in both groups received a regional block when possible, dexamethasone 8 mg at induction and paracetamol 1g plus dexketoprofen 50mg at the end of surgery. Continuous variables were compared using unpaired t-test (or Mann-Whitney U test) and categorical variables by Chi-square test. Statistical significance was set at p < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Patients who had Major Surgery for gynecologic cancers (cervix, endometrial, ovarian, vaginal, vulvar and breast cancer) under OFA and balanced anesthesia with opioids, both combined with regional anesthesia.

Exclusion Criteria:

* Patients who had Major Surgery for gynecologic cancers (cervix, endometrial, ovarian, vaginal, vulvar and breast cancer) under OFA and balanced anesthesia with opioids, but had later surgery with a different to previous anesthesia technique.
* Patients who had no later follow up during 12 months in the same Hospital, so we cannot register recurrence.

Ages: 20 Years to 91 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients who Major Surgery for gynecologic cancers (cervix, endometrial, ovarian, vaginal, vulvar and breast cancer)
Study Population: 132 women, aged 20-91 years old and ASA I-IV, who had Major Surgery for gynecologic cancers (cervix, endometrial, ovarian, vaginal, vulvar and breast cancer) under OFA and balanced anesthesia with opioids, both combined with regional anesthesia. They had surgery between February 2019 and February 2020 in Hospital La Paz de Madrid.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Systemic Inflammatory Response (C-Reactive Protein) | 48 hours after surgery
  To compare postoperative SIRS (Systemic Inflammatory Response) with C-Reactive Protein plasmatic level
Postoperative Systemic Inflammatory Response (Leucocytes Ratio) | 48 hours after surgery
  To compare postoperative SIRS (Systemic Inflammatory Response) with Leucocytes Ratio
Postoperative Systemic Inflammatory Response (Platelet Level) | 48 hours after surgery
  To compare postoperative SIRS (Systemic Inflammatory Response) with Platelet Level

SECONDARY OUTCOMES:
Time spent in the Post-Anesthesia Care Unit (PACU) | 30 days after surgery
  To compare recovery time between groups
Hospital stay | 30 days after surgery
  To compare hospital stay in both groups
Rate of later postoperative complications | 3 months after surgery
  Complications due to surgery which required hospitalization
Number of Participants with Cancer recurrence after surgery | 12 months after surgery
  To compare cancer recurrence (local and/or metastatic) 12 months after surgical treatment between groups.
Number of patients who Survive 12 months after surgery | 12 months after surgery
  To compare cancer survival 12 months after surgical treatment between groups

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Brogly, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Julia Albano Polo, Madrid, Spain

REFERENCES:
- [Background] Dubowitz JA, Sloan EK, Riedel BJ. Implicating anaesthesia and the perioperative period in cancer recurrence and metastasis. Clin Exp Metastasis. 2018 Apr;35(4):347-358. doi: 10.1007/s10585-017-9862-x. Epub 2017 Sep 11. PMID 28894976
- [Result] Malo-Manso A, Raigon-Ponferrada A, Diaz-Crespo J, Escalona-Belmonte JJ, Cruz-Manas J, Guerrero-Orriach JL. Opioid Free Anaesthesia and Cancer. Curr Pharm Des. 2019;25(28):3011-3019. doi: 10.2174/1381612825666190705183754. PMID 31298153
- [Result] Rossaint J, Zarbock A. Perioperative Inflammation and Its Modulation by Anesthetics. Anesth Analg. 2018 Mar;126(3):1058-1067. doi: 10.1213/ANE.0000000000002484. PMID 28922235
- [Result] Byrne K, Levins KJ, Buggy DJ. Can anesthetic-analgesic technique during primary cancer surgery affect recurrence or metastasis? Can J Anaesth. 2016 Feb;63(2):184-92. doi: 10.1007/s12630-015-0523-8. PMID 26497721
- [Result] Brown EN, Pavone KJ, Naranjo M. Multimodal General Anesthesia: Theory and Practice. Anesth Analg. 2018 Nov;127(5):1246-1258. doi: 10.1213/ANE.0000000000003668. PMID 30252709